CLINICAL TRIAL: NCT04561011
Title: Internet Delivered Cognitive Behavioural Therapy for Persons With Mild Traumatic Brain Injury: Pilot Phase 2
Brief Title: Internet Delivered Cognitive Behavioural Therapy for Persons With Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116271
Record Dates: First submitted 2020-09-01; First posted 2020-09-23 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-01

CONDITIONS: Mild Traumatic Brain Injury; Internet-Delivered Cognitive Behavioural Therapy; Depression; Anxiety
MeSH Terms: conditions — Brain Concussion; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants in will receive a guided online cognitive behaviour therapy program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons with Mild Traumatic Brain Injury (mTBI) (Experimental)
  Interventions: Behavioral: Internet-delivered Cognitive Behavioural Therapy(ICBT)

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioural Therapy(ICBT) — ICBT provides online structured self-help modules over several months based on the principles of CBT in combination with weekly guidance through emails and telephone calls. The course comprises 6 online lessons that provide psychoeducation about: 1) symptom identification and the cognitive behavioural model; 2) thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling; 4) graduated exposure/pacing; 5) memory and attention; and 6) relapse prevention. Participants will also have the opportunity to ask any questions regarding the content of the program materials and will receive a response from their Guide within 48-72 hours. Guide will spend ~15 mins. per week/per participant. All Guides have completed a university program (psychology or social work) and are registered clinicians or students working under supervision of a registered clinician.

SUMMARY:
Background: Individuals with neurological conditions (stemming from brain injury or stroke) can experience high levels of emotional distress leading to decreased quality of life and increased health care costs. Though mental health problems are prevalent and disabling, they often go untreated for various reasons, such as access to specialized care, rural and remote location, lack of time, or concerns about stigma related to seeking care. Internet delivered cognitive behaviour therapy (ICBT) overcomes barriers to face-to-face therapy by often reaching a much wider group of patients who experience unequal access to health care. The internet based program is based on cognitive behaviour therapy, which is an evidenced-based treatment that helps patients identify and modify thoughts and behaviours that contribute to their mental health concerns. ICBT has been shown to be effective in improving psychosocial outcomes such as depression and anxiety, along with disability and quality of life among persons with chronic health conditions.

Rationale: Despite evidence for ICBT among those with other chronic conditions, its efficacy has yet to be evaluated among those with neurological conditions such as brain injury and stroke.

Objective: The aim of the current study is to pilot an ICBT program developed through a patient oriented approach to improve overall wellbeing among those with mild traumatic brain injury.

Methods: In this project, an ICBT program for those with mild traumatic brain injury developed through an patient oriented approach (Phase 1) will be piloted amongst a small group of participants (n=20) to examine acceptability, feasibility, and limited efficacy. At the end of the program, participants will be asked to complete a brief semi-structured interview examining barriers and facilitators to the ICBT program. Participant feedback from the interviews will be used to further improve the ICBT program to meet the needs of the population. The results from the study will be used to guide larger studies to evaluate effectiveness of the program in a community setting.

Anticipated Impact: Ultimately, the proposed project aims to improve overall wellbeing and access to health care service for those who have mild traumatic brain injury and mental health concerns.

ELIGIBILITY:
Inclusion Criteria:

1. adults ≥ 18 years
2. diagnosed with mild traumatic brain injury (a neurological condition)
3. resident of Canada
4. access to a computer and the internet
5. cognitive capacity to read and understand the content of the program.

Exclusion Criteria:

1. High risk of suicide
2. Serious cognitive impairment or dementia (<21 on the Telephone Interview of Cognitive Status (TICS)
3. primary problems with psychosis, alcohol or drug problems, mania
4. Currently receiving active psychological treatment for anxiety or depression
5. Not present in Canada during treatment; 6) Concerns about online therapy
6. Physically unable to perform the tasks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Change in depression | Baseline to 3 months.
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27.

SECONDARY OUTCOMES:
Change in anxiety | Baseline to 3 months.
  Generalize Anxiety Disorder - 7 Item (GAD7). Higher total scores indicate greater severity of anxiety. Scores range from 0 to 21.
Change in quality of life | Baseline to 3 months.
  EuroQol five-dimension (EQ-5D) questionnaire. Every dimension of the EQ-5D-5L includes five answer levels, covering no problems (1) to extreme problems (5). Higher numbers indicates poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Swati Mehta, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Josephs Parkwood Institute, London, Ontario, Canada